CLINICAL TRIAL: NCT02405260
Title: A Multi-Center, Adaptive Phase 2, Randomized, Double-Blind, Placebo- and Active-Controlled (Sitagliptin), Parallel Group Study to Evaluate the Safety and Efficacy of TTP399 Following 6 Months Administration in Subjects With Type 2 Diabetes Mellitus on A Stable Dose of Metformin
Brief Title: Add Glucokinase Activator to Target A1c
Acronym: AGATA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTP399-202
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TTP399; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TTP399 400 mg (Experimental): TTP399 once daily
  Interventions: Drug: TTP399 400 mg
- TTP399 800 mg (Experimental): TTP399 once daily
  Interventions: Drug: TTP399 800 mg
- Sitagliptin 100 mg (Active Comparator): Sitagliptin once daily
  Interventions: Drug: Sitagliptin 100 mg
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTP399 400 mg — once daily
  Arms: TTP399 400 mg
Drug: TTP399 800 mg — once daily
  Arms: TTP399 800 mg
Drug: Sitagliptin 100 mg — once daily
  Arms: Sitagliptin 100 mg
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
This trial is a multi-center, adaptive, randomized, double-blind, placebo- and active- controlled, parallel group, Phase 2 study in subjects with T2DM to evaluate the effect of TTP399 on HbA1c following administration for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* A historical diagnosis of Type 2 Diabetes in accordance with the American Diabetes Association (ADA) guidelines, with diagnosis at least 6 months prior to Screening.
* On a stable (for the last 3 months prior to screening) regimen of metformin monotherapy equivalent of at least 1000 mg once daily.
* Males, females of childbearing potential (must have a negative pregnancy test and be willing to comply with protocol contraception), and females of non-childbearing potential.
* Age 18 to 75 years, inclusive, at the time of screening.
* HbA1c ≥7.0% and ≤9.5%.
* Generally stable health without active infection or history of major surgery or significant injuries within the last year.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus, maturity-onset diabetes of the young, insulin-requiring Type 2 Diabetes, other unusual or rare forms of diabetes mellitus, or history of diabetic ketoacidosis.
* Clinically significant abnormal lab values including eGFR <50ml/min/1.73m2, ALT, bilirubin or AST >1.5 X ULN, hypokalemia or other clinically significant electrolyte abnormality.
* History of myocardial infarction, unstable angina, coronary revascularization, stroke, or transient ischemic attack within 2 years of screening.
* Presence of symptomatic congestive heart failure.
* History of cardiac arrhythmias requiring treatment or prophylaxis with drugs or devices during the last 2 years or any history of atrial fibrillation or flutter beyond a single short-term episode (e.g., lasting 1-2 days).
* History or presence of a 2nd degree or greater atrioventricular block in the absence of a pacemaker.
* A 12-lead ECG, from screening or baseline demonstrating QTcF interval >450 msec for males or >47 msec for females.
* A family or personal history of long QT syndrome.
* History of pancreatitis.
* Persistent, uncontrolled hypertension.
* Presence of chronic active hepatitis (hepatitis B, hepatitis C, nonalcoholic steatohepatitis [NASH]) and/or known liver cirrhosis.
* Participation in any formal weight loss program, or fluctuation of > 5% in body weight, or having received medications approved for weight loss within 3 months prior to screening.
* A positive pre-study drug screen.
* Participation in a clinical trial and receipt of an investigational product within 30 days.
* Have a history of drug abuse within 2 years of screening or a positive pre-screen drug screen.
* Have a history of hypoglycemic episode requiring glucose, glucagon, or orange juice administered by someone other than the patient within 6 months prior to screening.
* A history of excessive alcohol consumption within the last 2 years prior to screening
* Mental or legal incapacitation.
* Blood donation of approximately 1 pint (500 mL) within 8 weeks.
* History of MEN-2 or family history of medullary thyroid cancer.
* History of cancer, other than non-melanoma skin cancer, that required therapy in the 5 years prior study start.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (Glycosylated haemoglobin) | Day 1 to Day 168

SECONDARY OUTCOMES:
HbA1c < 7% at 6 months | Day 1 to Day 168
HbA1c < 6.5% at 6 months | Day 1 to Day 168
Plasma Glucose Levels | Day 1 to Day 168
Lipid Levels | Day 1 to Day 168
Insulin Levels | Day 1 to Day 168
Lactate Levels | Day 1 to Day 168
C-peptide Levels | Day 1 to Day 168
Glucagon Levels | Day 1 to Day 168
Glucagon-like Peptide-1 Levels | Day 1 to Day 168
Change in Body Weight | Day 1 to Day 168
Adverse Events | Day 1 to Day 182
Blood Pressure | Day 1 to Day 182
Electrocardiogram Parameters | Day 1 to Day 182
Hematology | Day 1 to Day 182
Blood Chemistry | Day 1 to Day 182
Urinalysis | Day 1 to Day 182
Pulse | Day 1 to Day 182

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Valcarce, Ph.D., Study Chair — vTv Therapeutics
Locations (19):
- United States (19):
  - Mesa, Arizona
  - Tuscon, Arizona
  - Canoga Park, California
  - Huntington Park, California
  - Los Angeles, California
  - West Hills, California
  - Centennial, Colorado
  - Littleton, Colorado
  - Waterbury, Connecticut
  - West Palm Beach, Florida
  - Gurnee, Illinois
  - Evansville, Indiana
  - Rochester, Minnesota
  - Greensboro, North Carolina
  - Moncks Corner, South Carolina
  - San Antonio, Texas
  - Schertz, Texas
  - Norfolk, Virginia
  - Richland, Washington